CLINICAL TRIAL: NCT05749575
Title: A Prospective, Open-label, Phase II Clinical Trial of Chidamide, PD-1 Monoclonal Antibody and Paclitaxel in Neoadjuvant Therapy for Low Hormone Receptor(HR) Expression,HER2-negative Early Breast Cancer.
Brief Title: Chidamide Plus PD-1 Plus Paclitaxel of Neoadjuvant Treatment in Low HR Expression,HER2-negative Early Breast Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Associate Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-2022-02
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; toripalimab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide Plus Toripalimab Plus Paclitaxel (Experimental): Cedaramine: 20mg, twice a week.Toripalimab: 240mg, once in 3 weeks,intravenous.Paclitaxel: 175mg / m2, once in 3 weeks, routine preventive anti-allergy treatment, surgery after 4 cycles of IV infusion.
  Interventions: Drug: Chidamide Plus Toripalimab Plus Paclitaxel

INTERVENTIONS:
Drug: Chidamide Plus Toripalimab Plus Paclitaxel — Each participant receives chidamide plus toripalimab plus paclitaxel

SUMMARY:
Triple-negative breast cancer has always been a difficult problem in clinical practice because of its young onset age, high aggressiveness, no clear therapeutic target and poor clinical prognosis. The treatment of triple-negative breast cancer is mainly chemotherapy, and in order to break the current dilemma, new treatments must be introduced. Immunotherapy is one of the most high-profile treatments. The KEYNOTE-522 study and Impassion 031 Study have found that immunotherapy can significantly improve the pCR of patients with triple yin breast cancer, rate, independent of PD-L1 expression status, and good safety.Cedardenamine is a histone deacetylation (HDAC) inhibitor developed in China.Many studies suggest that the use of sidabamine will likely enhance the efficacy of PD-1 / PD-L1 mAb in breast cancer and expand the use of PD-1 / PD-L1 mAb in the beneficiary population of breast cancer

DETAILED DESCRIPTION:
Cedaramine can effectively inhibit subtypes 1,2,3 of HDAC class I and type 10 of class IIb. Sidabamide can directly induce cycle arrest and apoptosis in tumors and has demonstrated its clinical role in lymphoma and breast cancer.besides, In recent years, many studies have found that HDAC inhibitors also have their functions in regulating immunity, Such as: 1) upregulated tumor antigen / co-stimulatory molecule / receptor levels of tumor cells (such as MHC I / II, PRAME, MIC A/B, PDL-1, etc.), Make it easier to be recognized by the immune system; 2) Initialize the natural immune system, Activating NK cell activity; 3) Initialize the acquired immune system, Activating initial T cells (Naive T cells) to target tumor antigen; 4) Increase the CD8 + effector cells that kill tumor cells, Downregulation of the immunosuppressive cells, Such as the Treg 6 7 and MDSC, Promote the formation and maintenance of acquired immune memory T cells. Preclinical studies suggested that HDAC was synergistic with PD-1 / PD-L1 antibodies and could serve as a sensitizer for PD-1 / PD-L1 antibodies. A phase I study in solid tumors found that sitabenamine combined with natureumab had an objective response rate (ORR) of 48% and a disease control rate (DCR) of 87%.Therefore, we conduct this study to observe the efficacy and safety of neoadjuvant therapy in early HR low-expression ,HER2-negative breast cancer patients treated with PD-1 mAb and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1.18-75 years old. 2.ECOG whole-body status (performance status , PS) grade 0 to 1. 3.ER and PR IHC showed <10% staining and HER2 negative. 4.The patients who receive at least 2 neoadjuvant sessions with anthracycline are assessed to SD (4 anthracycline-containing sessions) or PD with breast MRI, CT or ultrasound according to the RECIST standard.

5.The patients refuse prior surgical treatment (the patient requires breast preservation, but it cannot be performed by surgical consultation), or it is not suitable for prior surgical treatment.

6.The main organ function is normal, that is, to meet the following criteria:

1. the criteria for blood routine examination:

   1. ANC≥1.5×109/L；
   2. PLT≥100×109/L；
   3. Hb≥90g/L；
2. the criteria for biochemical examination:

   1. TBIL<1.5×ULN；
   2. ALT and AST<2.5×ULN；
   3. BUN and Cr ≤ 1.5 × ULN or endogenous creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault formula).

      7.No malabsorption or other gastrointestinal disorders that affect drug absorption 8.Serum pregnancy tests for women of childbearing age must be negative within 7 days before treatment; all enrolled patients (whether male or female) should have adequate barrier contraception throughout the treatment period and within 4 weeks of treatment.

      9.The subjects volunteer to join the study and sign informed consent, with good compliance and cooperated with follow-up.

      Exclusion Criteria:
      1. Previous use of investigational drugs such as PD-1 or PD-L1 mAb; sidabamine or other HDAC inhibitors, and taxane-based chemotherapies (including paclitaxel or docetaxel).
      2. Distant metastases, but enrollment could be considered if the distant metastatic lesion is confined to the ipsilateral cervical lymph exclusion criteria node only.
      3. Unstable systemic disease (including active infection, poorly controlled hypertension, unstable angina pectoris, congestive heart failure, hepatic, renal, or metabolic disease, etc).
      4. Any other malignancy within five years (except completely cured cervical carcinoma in situ or basal or squamous epithelial skin carcinoma).
      5. For known human immunodeficiency virus (HIV) infection, hepatitis B virus carriers must be treated for anti-hepatitis B virus replication during antitumor therapy.
      6. Prior history of clear neurological or psychiatric disorders, including epilepsy or dementia.
      7. Pregnant or lactating women.
      8. Any unstable or potentially jeopardizing patient safety and its compliance to the study.
      9. Other situations that investigators think it is unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Pathology tpCR (ypT0/is, ypN0) rate | 1 year
  After completion of neoadjuvant therapy and surgery, there was no residual invasive carcinoma in the pathological evaluation of hematoxylin-and eosin-stained resected breast cancer samples and all ipsilateral lymph node samples. Count pCR rate in patients undergoing surgery.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  The proportion of subjects who achieved CR or PR as optimal tumor response in the ITT population, as assessed by the efficacy evaluation criteria for solid tumors (RECIST1.1).
Disease-free survival (DFS) | 1 year
  Defined as the time interval from the first day of no disease (the date of surgery) to the first recording of a related event, including postoperative disease recurrence or metastasis and death from any cause.
Disease-free survival in 3 years | 3 year
  Defined as disease-free survival for all patients undergoing surgery from the first day of no disease ( the date of surgery) to 3 years.
Event-free survival (EFS) | 1 year
  Defined as the time interval from the first day of no disease (the date of surgery) to the first recording of related events, including postoperative disease recurrence or metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No